CLINICAL TRIAL: NCT05995782
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, SAD and MAD Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral FB418 in Healthy Adult Subjects and Healthy Elderly Subjects
Brief Title: A Phase 1, SAD and MAD Study to Evaluate the Safety and Tolerability of FB418
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: 1ST Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FB418_P101
Record Dates: First submitted 2023-08-07; First posted 2023-08-16 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease Psychosis; Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FB418 (Experimental): Part A - Single ascending oral doses of FB418 in healthy adult subjects and healthy elderly subjects.
  Part B - Multiple ascending oral doses FB418 in healthy adult subjects.
  Interventions: Drug: FB418
- FB418-Placebo (Placebo Comparator): Part A - Single Ascending Dose matching placebo study Part B - Multiple Ascending Dose matching placebo study
  Interventions: Drug: FB418

INTERVENTIONS:
Drug: FB418 — Oral dose
  Other Names: FB418 active drug

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics and pharmacodynamics of oral doses of FB418 in healthy adult subjects and healthy elderly subjects.

DETAILED DESCRIPTION:
Part A:

Primary:

To assess the safety and tolerability of single ascending oral doses of FB418 in healthy adult subjects and healthy elderly subjects.

Secondary:

To assess the pharmacokinetics (PK) of FB418 and metabolite after single ascending oral doses of FB418 in healthy adult subjects and healthy elderly subjects.

To assess the effect of a high-fat meal on the PK of FB418 and metabolite after a single oral dose of FB418 when administered to healthy adult subjects.

Part B:

Primary:

To assess the safety and tolerability of multiple ascending oral doses FB418 in healthy adult subjects.

Secondary:

To assess the PK of FB418 and metabolite after multiple ascending oral doses of FB418 in healthy adult subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy, adult, male 19 55 years of age, inclusive, at the screening.
2. For elderly subjects(Part A Cohort 5 only), healthy, elderly, male or female (of non childbearing potential only) over 60 years of age, inclusive, at screening.
3. In the case of the elderly(Part A Cohort 5 only), they have a history of mild disease, but can participate if the researcher judges that they can stop taking the drug at least 2 weeks before the expected first dose or before the half-life is 5 times or more)
4. The continuous non smoker who have not used nicotine containing products for at least 3 months prior to (the first) dosing and throughout the study are based on subjective self reporting.
5. Body mass index (BMI) ≥ 18 and ≤ 32 kg/m2 at the screening.
6. Medically healthy with no clinically significant medical history, physical examination, simplified neurological examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
7. In Cohort 5, A female subject must be of non childbearing potential

Key Exclusion Criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of a clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. Is at suicidal risk in the opinion of the PI as per the following criteria:

   1. Any suicide attempts within 12 months prior to screening or any suicidal intent, including a plan, within 3 months prior to screening.
   2. C-SSRS answer of "YES" on suicidal ideation within 3 months prior to screening.
5. History or presence of alcoholism or drug abuse within the past 2 years prior to (the first) dosing.
6. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
7. History of seizures (childhood febrile seizures are excepted).
8. Positive urine drug or alcohol results at screening or check in.
9. Has an abnormal screening ECG indicating a second- or third- degree AV block, or one or more of the following: QRS > 120 msec, QTcF > 450 msec for males and > 460 msec for females, PR interval > 220 msec. Any rhythm other than normal sinus rhythm, which is interpreted by the PI or designee to be clinically significant at screening or check-in.
10. Has any medical or surgical condition in which lumbar puncture is contraindicated in the opinion of the PI.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events (TEAE) | Up to 7 ~ 14 days after the last dose
  Number of TEAEs including serious adverse events (SAEs)

SECONDARY OUTCOMES:
PK parameter 1 | Up to 72 hours after the last dose
  Maximum observed concentration (Cmax) of FB418 in plasma
PK parameter 2 | Up to 72 hours after the last dose
  Time to maximum observed concentration (Tmax) of FB418 in plasma
PK parameter 3 | Up to 72 hours after the last dose
  The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of FB418 in plasma
PK parameter 4 | Up to 72 hours after the last dose
  Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) of FB418 in plasma
PK parameter 5 | Up to 72 hours after the last dose
  Apparent terminal elimination half-life (t1/2) of FB418 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: 1STBIO study manager, Study Director — 1ST Biotherapeutics, Inc.
Locations (1):
- Seoul National University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No